CLINICAL TRIAL: NCT01274026
Title: Evaluation of Behavior, Executive Function, Neurotransmitter Function and Genomic Expression in PKU "Nonresponders" to Kuvan® (Sapropterin Dihydrochloride)
Brief Title: Evaluation of Behavior, Executive Function, Neurotransmitter Function and Genomic Expression Kuvan Nonresponders
Acronym: IST
Status: Completed | Type: Observational
Sponsor: Tulane University School of Medicine (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Other Study IDs: 183590-1
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Phenylketonuria; Behavior and Behavior Mechanisms; PAH Gene Expression
Keywords: phenylketonuria; PKU; phenylalanine; neurotransmitters; gene; Kuvan; sapropterin
MeSH Terms: conditions — Phenylketonurias; Behavior | interventions — sapropterin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- evaluation of benefit of sapropterin: Intervention 'sapropterin dihydrochloride': 20 individuals, either known to be non-responsive, or naive to sapropterin, are given a 4 week administration of sapropterin. Pre-, and Post- evaluation of behavior, executive function, neurotransmitter function, and genomic expression are assessed and evaluated for change.
  Interventions: Drug: sapropterin dihydrochloride

INTERVENTIONS:
Drug: sapropterin dihydrochloride — In 30 PKU patients found previously to exhibit no decrease in blood PHE levels behavioral and cognitive function, neurotransmitter levels, and gene expression of enzyme activity will be measured at baseline and after 4 weeks of Kuvan administration. Rating inventories of executive function performance and behavior will be administered to patients and parents.
  Urine neurotransmitters, blood microarray expression, and plasma amino acids will be measured (plasma PHE and TYR levels will also be measured at weeks 1 and 2). Nutrient analysis of 3 day food diaries will be conducted.
  Other Names: Kuvan

SUMMARY:
This observational study seeks to establish evidence:

1. that physiologic changes, unrelated to effect on the Phenylalanine Hydroxylase (PAH) enzyme, occur in Phenylketonuria (PKU) patients who are treated with sapropterin (Kuvan®) therapy,
2. that these changes may be caused by enhanced neurotransmitter synthesis in the brain or an upregulation of gene expression (increasing the ability of genes to produce functional enzymes),
3. and that beneficial changes in behavior and cognition, especially executive functioning skills may result.

The objective of this study is to correlate any change in behavior and executive function skills of PKU patients who are non-responsive to sapropterin effect on the PAH enzyme, as defined by lowered blood PHE levels, with urine neurotransmitter levels and broad gene expression prior to and after sapropterin administration.

Expected outcomes would include evidence of sapropterin effects on upregulation of enzymes other than PAH that control neurotransmitter synthesis, and any resulting correlation with behavioral and cognitive changes.

The investigators hope this study will inform further detailed investigations into the biochemical and molecular actions of sapropterin (Kuvan®) that lead to increased understanding of possible treatment effects beyond a lowered blood PHE response.

DETAILED DESCRIPTION:
The anticipated study participant population was approximately 30 established PKU patients receiving care from Hayward Genetics Center, who were found previously to exhibit no decrease in blood phenylalanine (PHE) levels (nonresponders) with administration of sapropterin. Subjects acted as their own controls. An additional number of patients naive to sapropterin were subsequently added to the study, and the age exclusion of over 21 years of age was omitted per IRB approval. Primary endpoints were designed to be measurement of behavioral and cognitive function, neurotransmitter levels, and gene expression of enzyme activity after 4 weeks on treatment compared to baseline levels.

At study baseline each patient attended an approximately 1 hour clinic visit at their usual genetics clinic location. Study purpose, design, and requirements were discussed, and consents/assents reviewed and signed.

Rating inventories of executive function performance and behavior (BASC-2 and BRIEF tools) were administered to patients and parents by the Principal Investigator (PI) and/or the Study Coordinator.

Urine samples were collected non-invasively for measurement of neurotransmitter levels. Blood as collected by venipuncture (3-5 ml) for microarray expression analysis and analysis of plasma amino acids. 3-day food records previously provided to participants for completion were collected.

Participants were provided with a 4 week supply of Kuvan® and instructions on how to take the medication during the study period. The importance of maintaining usual dietary intake (food choices and metabolic formula) to minimize any research effect not attributable to sapropterin administration was emphasized. Sapropterin was discontinued at the end of the 4 week study period. The exception to this was for the naive patients who were found to be responsive to sapropterin.

All of these measures were repeated at the same sites with study participants at the end of week 4 of the study period.

At the ends of weeks 1 and 2 additional blood samples were sent to Hayward Genetics Center for measurement of PHE and tyrosine (TYR) levels to ascertain no significant changes have occurred in a patient's usual dietary intake. These samples were drawn at each patient's local state health unit, as is done for usual monitoring. Nutrient analysis of the 3-day food diaries was conducted at Hayward Genetics Center.

1. Behavior and executive function were assessed using published validated inventories, completed as patient self-reports and as parent (or guardian) reports when appropriate. Instruments used were the Behavioral Assessment System for Children (BASC-2) parental Rating Scale and Self-Reporting Personality Rating Scale, and the Behavioral Rating Inventory of Executive Function (BRIEF) Parent Form Instruments of Executive Function. Completed inventories were scored using electronic evaluation instruments by the Study Coordinator and PI, with consultation from Harvard Medical Center experts as needed.
2. Urine samples were non-invasively collected and sent for analysis of catechols and neurotransmitters to an NIH laboratory specializing in this technique. Samples were blinded to this laboratory to prevent bias.
3. Microarray analysis of blood samples was conducted at Hayward Genetics Molecular Laboratory to determine any effect on gene expression, and thus enzyme activity, as a result of sapropterin administration.
4. Plasma amino acids were analyzed at Hayward Genetics Biochemical Laboratory to document that patients are "nonresponsive" to sapropterin (no resultant lowering of blood PHE); and to monitor any changes in plasma amino acids that could indicate a patient's failure to maintain usual dietary restrictions. Patients naive to Kuvan who responded were noted and function as comparators.
5. 3-day food diaries completed by patients (or parent/guardians) at home documented any substantive changes in usual dietary intake during the study period. These were analyzed at Hayward Genetics Center using the MetabolicPro web-based analysis program.

ELIGIBILITY:
Inclusion Criteria:

* established Hayward Genetics Center patients:
* confirmed diagnosis of PKU,
* aged 2-21 years,
* not responsive to sapropterin with decreased blood PHE levels Subsequent to the start of the study inclusion criteria were amended: the upper limit of age was omitted, and a limited number of patients who were naive to sapropterin were recruited.

Exclusion Criteria:

* pregnancy
* preexisting cognitive disorder or concurrent disease that would interfere with participation,
* documented equal to or greater than 20% decrease in blood PHE levels as a response to sapropterin administration,
* receiving neurotransmitter supplementation or medication for attention deficit hyperactivity disorder (ADHD),
* received sapropterin therapy in the 2 months prior to the study

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study participants were solicited from treated patients diagnosed with PKU who are followed by our clinic. Participants were initially limited to those who had undergone a trial with sapropterin (FDA approved drug available for treatment) as part of their clinical care and been found to be non-responsive. Subsequently, with IRB approval, some patients diagnosed with PKU from our clinic population who were naive to sapropterin were added to the study.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in behavior as a result of Kuvan administration | assessment during a 4 week trial of Kuvan
  This study seeks to establish evidence that behavioral changes, unrelated to blood phenylalanine levels, occur in PKU patients who are treated with Kuvan therapy, and that beneficial changes in behavior as measured by validated measurement questionnaires may result.
change in executive function as a result of Kuvan administration | assessment during a 4 week trial of Kuvan
  This study seeks to establish evidence: that cognitive changes unrelated to blood phenylalanine levels occur in PKU patients who are treated with Kuvan therapy, and that beneficial changes in cognition, especially executive functioning skills as measured by validated measurement questionnaires may result.

SECONDARY OUTCOMES:
change in neurotransmitter synthesis | assessment during a 4 week trial of Kuvan administration
  This study seeks to establish evidence:
  that physiologic changes, unrelated to effect on the PAH enzyme, occur in PKU patients who are treated with Kuvan® therapy,and that these changes may be caused by enhanced neurotransmitter synthesis in the brain or an upregulation of gene expression (increasing the ability of genes to produce functional enzymes), Expected outcomes would include evidence of sapropterin effects on upregulation of enzymes other than PAH that control neurotransmitter synthesis, and any resulting correlation with behavioral and cognitive changes.

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Andersson, MD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University Health Science Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No